CLINICAL TRIAL: NCT01476215
Title: A Pharmacokinetic Study Investigating the Rate and Extent of Paracetamol Absorption of Three Experimental Sustained Release Pediatric Suspensions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3950669
Record Dates: First submitted 2011-11-03; First posted 2011-11-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: paracetamol
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fast dissolution suspension (Experimental)
  Interventions: Drug: Paracetamol fast dissolution suspension
- Medium dissolution suspension (Experimental)
  Interventions: Drug: Paracetamol medium dissolution suspension
- Slow dissolution suspension (Experimental)
  Interventions: Drug: Paracetamol slow dissolution suspension
- Marketed suspension (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol fast dissolution suspension
  Arms: Fast dissolution suspension
Drug: Paracetamol medium dissolution suspension
  Arms: Medium dissolution suspension
Drug: Paracetamol slow dissolution suspension
  Arms: Slow dissolution suspension
Drug: Paracetamol
  Arms: Marketed suspension

SUMMARY:
This proof of principle PK study will allow GSKCH to select the most favorable sustained release formulation among 3 prototypes to move to the next stage of drug development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Body Mass Index between 19.0 - 28.0 (kg/m2) inclusive

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Time to plasma level above therapeutic level | baseline to 8 hours

SECONDARY OUTCOMES:
General PK parameters (e.g. AUC, Tmax, Cmax) | baseline to 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services NEBRASKA, Lincoln, Nebraska, United States